CLINICAL TRIAL: NCT02532894
Title: Effects of E-smoke on Levels of Endothelial Progenitor Cells and Microparticles in Healthy Volunteers
Acronym: ESMOKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Magnus Lundbäck, MD, PhD,, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 214/552-31/4
Record Dates: First submitted 2015-08-24; First posted 2015-08-26 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Healthy
Keywords: endothelial dysfunction; microvesicles; endothelial progenitor cells; electronic cigarettes
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esmoke (Experimental): Inhaling e-cigarette vapor
  Interventions: Device: Electronic cigarette
- Control (No Intervention)

INTERVENTIONS:
Device: Electronic cigarette — Inhaling e-cigarette vapor
  Arms: Esmoke

SUMMARY:
We plan to investigate the acute effects of inhaling e-cigarette vapor on cell function measured by microvesicles and endothelial progenitor cells. Micro vesicles are released upon either activation or apoptosis from different cell types such as platelets, leucocytes and endothelial cell. Endothelial progenitor cells are a type of stem cells that circulate in the blood with the ability to differentiate to endothelial cells. Endothelial progenitor cells are inversely correlated to cardiovascular risk factors.

As a secondary endpoint we plan to investigate exhaled nitric oxide - a common inflammation marker used in asthmatic patients - after inhalation of electronic cigarette vapor.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* sporadic cigarette smoking (<9 cigarettes per month)

Exclusion Criteria:

* Any form of cardiovascular disease
* Any form of pulmonary disease like asthma or COPD
* Any form of systemic or chronic disorder like rheumatologic or metabolic diseases.
* Active allergy within 4 weeks of the study
* Symptoms of infection or inflammation within 4 weeks of the study
* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10; Primary Completion 2014-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in number of endothelial progenitor cells | 24 hours
Change in number of micro vesicles | 24 hours

SECONDARY OUTCOMES:
Change in exhaled nitric oxide | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Lundbäck, MD, PhD, Principal Investigator — Institutionen för kliniska vetenskaper, Danderyds sjukhus
Locations (1):
- Institutionen för kliniska vetenskaper, Danderyds sjukhus, Danderyd, Stockholm County, Sweden